CLINICAL TRIAL: NCT02607228
Title: A Phase 1b/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GS-5829 as a Single Agent and In Combination With Enzalutamide in Subjects With Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GS-5829 (Alobresib) as a Single Agent and In Combination With Enzalutamide in Participants With Metastatic Castrate-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-350-1604; 2015-003741-26 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Castrate-Resistant Prostate Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Alobresib Dose Escalation (Experimental): Participants who have progressed on either abiraterone and/or enzalutamide will be enrolled to receive increasing doses of alobresib up to 9 mg to determine the MTD.
  Interventions: Drug: Alobresib
- Alobresib + Enzalutamide Dose Escalation (Experimental): Following a two week lead-in with enzalutamide once daily, participants who have progressed on abiraterone will receive less than or equal to MTD of alobresib in combination with enzalutamide 160 mg once daily. Based on observed pharmacokinetics (PK) interaction, toxicity, and tolerability observed in the single agent dose escalation, the dose of alobresib may be increased.
  Interventions: Drug: Alobresib; Drug: Enzalutamide
- Alobresib Dose Expansion (Group 1) (Experimental): Participants will receive a dose less than or equal to MTD of alobresib (based on safety, pharmacodynamics (PD), and tolerability).
  Interventions: Drug: Alobresib
- Alobresib + Enzalutamide Dose Expansion (Group 2) (Experimental): Participants will receive a dose less than or equal to MTD of alobresib plus enzalutamide (based on safety, PD, and tolerability).
  Interventions: Drug: Alobresib; Drug: Enzalutamide
- Alobresib + Enzalutamide Dose Expansion (Group 3) (Experimental): Participants will receive alobresib plus enzalutamide (dose will be equivalent to the dose chosen for Group 2).
  Interventions: Drug: Alobresib; Drug: Enzalutamide

INTERVENTIONS:
Drug: Alobresib — Tablet administered orally once daily.
  Other Names: GS-5829
Drug: Enzalutamide — Capsules administered orally once daily.
  Other Names: XTANDI®
  Arms: Alobresib + Enzalutamide Dose Escalation; Alobresib + Enzalutamide Dose Expansion (Group 2); Alobresib + Enzalutamide Dose Expansion (Group 3)

SUMMARY:
This study consists of two phases: Dose Escalation (Phase 1b) and Dose Expansion (Phase 2)

The Dose Escalation phase will characterize the safety, tolerability, and determine the maximum tolerated dose (MTD) of alobresib as a single agent and in combination with enzalutamide, in participants with metastatic castrate-resistant prostate cancer (mCRPC).

The Dose Expansion phase will evaluate the following:

* In group 1, the efficacy of alobresib as a single agent in participants with mCRPC who have progressed while receiving enzalutamide (may have also received abiraterone)
* In group 2, the efficacy of alobresib combined with enzalutamide in participants with mCRPC who have progressed while receiving treatment with abiraterone (may not have previously received enzalutamide)
* In group 3, the efficacy of alobresib combined with enzalutamide in participants with mCRPC who have had prostate specific antigen (PSA) progression, but not radiographic progression, while receiving treatment with enzalutamide (participants may have also previously received abiraterone)

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer (individuals with primary neuroendocrine carcinoma of prostate are excluded)
* Must have documented progressive disease by meeting at least one of the Prostate Cancer Working Group 2 Criteria
* Castration resistant disease defined as ongoing androgen deprivation therapy with gonadotropin-releasing hormone (GnRH) analogue or bilateral orchiectomy and serum testosterone level ≤ 1.73 nmol/l (50 ng/dL) at screening visit. Individuals who have not had a bilateral orchiectomy must have a plan to maintain effective GnRH-analogue therapy for the duration of the trial.
* Metastatic disease documented by bone lesions on bone scan or by measurable soft tissue disease by computerized tomography/magnetic resonance imaging (CT/MRI). Patients whose disease spread is limited to regional pelvic lymph nodes are not eligible
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* Adequate organ function defined as follows:

  * Hematologic: Platelets ≥ 100 x 10^9/L; Hemoglobin ≥ 9.0 g/dL; absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (without platelet transfusion or any growth factors within previous 7 days of the hematologic laboratory values obtained at screening visit)
  * Hepatic: Aspartate transaminase (AST) / Alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN) (if liver metastases are present, ≤ 5 x ULN); Total or conjugated bilirubin ≤ 1.5 x ULN
  * Renal: Serum Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 60 mL/min as calculated by the Cockroft-Gault method
* Coagulation: International Normalized Ratio (INR) ≤ 1.2

Key Exclusion Criteria:

* Known brain metastasis or leptomeningeal disease
* Myocardial infarction, symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, or serious uncontrolled cardiac arrhythmia within the last 6 months of Cycle 1 Day 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of alobresib, including any unresolved nausea, vomiting, or diarrhea that is Common Terminology Criteria for Adverse Events (CTCAE) Grade > 1
* Anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy) within 21 days or 5 half-lives, whichever is longer, of study drug dosing (6 weeks for nitrosoureas, mitomycin C, or molecular agents with t1/2 > 10 days); concurrent use of an luteinizing hormone releasing hormone (LHRH) agonist is permitted for all individuals and ongoing enzalutamide is required in Group 3.
* History of long QT syndrome or whose corrected QT interval (QTc) measured (Fridericia method) at screening is prolonged (> 450 ms).
* Prior exposure to bromodomain (BET) inhibitors
* Clinically significant bleeding within 28 days of Cycle 1 Day 1
* Known human immunodeficiency virus (HIV) infection
* Hepatitis B surface antigen (HBsAg) positive
* Hepatitis C virus (HCV) antibody positive
* Use of moderate/strong cytochrome P450 (CYP)3A4 inhibitors or moderate/strong CYP3A4 inducers within 2 weeks prior to the first dose of study drug (with the exception of enzalutamide in the combination arms)
* Evidence of bleeding diathesis
* History of hemoptysis of ≥ 2.5 mL/1 teaspoon within 6 months of Cycle 1 Day 1
* History of high grade esophageal or gastric varices
* Anticoagulation/antiplatelet therapy within 7 days of Cycle 1 Day 1, including low molecular weight heparin, or warfarin.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- United States (4):
  - San Francisco, California
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 4 study sites in the United States. The first participant was screened on 08 December 2015. The last study visit occurred on 03 September 2019. Phase 2 Dose Expansion of the study was not conducted. Results are reported for only Dose Escalation Monotherapy and Combination Therapy.
Pre-assignment Details: 43 participants were screened.
Groups:
- Monotherapy: Alobresib 2 mg: Participants who had progressed on either abiraterone and/or enzalutamide, received alobresib 2 mg tablets administered orally once daily to determine the maximum tolerated dose (MTD).
- Monotherapy: Alobresib 3 mg: Participants who had progressed on either abiraterone and/or enzalutamide, received alobresib 3 mg tablets administered orally once daily to determine the MTD.
- Monotherapy: Alobresib 4 mg: Participants who had progressed on either abiraterone and/or enzalutamide, received alobresib 4 mg tablets administered orally once daily to determine the MTD.
- Monotherapy: Alobresib 6 mg: Participants who had progressed on either abiraterone and/or enzalutamide, received alobresib 6 mg tablets administered orally once daily to determine the MTD.
- Monotherapy: Alobresib 9 mg: Participants who had progressed on either abiraterone and/or enzalutamide, received alobresib 9 mg tablets administered orally once daily to determine the MTD.
- Combination Therapy: Alobresib 3 mg + Enzalutamide: Participants who had progressed on abiraterone, received alobresib 3 mg tablets administered orally once daily in combination with enzalutamide 160 mg capsules administered orally once daily.
- Combination Therapy: Alobresib 6 mg + Enzalutamide: Participants who had progressed on abiraterone, received alobresib 6 mg tablets administered orally once daily in combination with enzalutamide 160 mg capsules administered orally once daily.
Period: Overall Study
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Started | 5 | 4 | 3 | 6 | 5 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 4 | 3 | 6 | 5 | 6 | 2
Not completed — Progressive Disease | 4 | 3 | 1 | 5 | 4 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 1 | 1 | 1
Not completed — Investigator's Discretion | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrew Consent | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Analysis Set included all participants who received a study participant identification number in the study after screening.
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide | Total
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 6 | 2 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (9.28) | 67.3 (10.69) | 67.7 (5.69) | 66.8 (9.39) | 69.2 (6.61) | 62.5 (10.23) | 67.0 (0.00) | 66.7 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 4 | 3 | 6 | 5 | 6 | 2 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 5 | 4 | 3 | 6 | 3 | 5 | 2 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Race: White | 4 | 4 | 2 | 6 | 4 | 5 | 2 | 27
  Race: Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 3 | 6 | 5 | 6 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b Dose Escalation: Number of Participants Experienced Dose Limiting Toxicities (DLTs)
Description: A DLT was a toxicity, considered possibly related to alobresib, and which occurred during the DLT assessment window (Days 1 through 28) in each cohort: Grade ≥ 4 neutropenia (absolute neutrophil count (ANC) < 500/mm^3), Grade ≥ 3 neutropenia (ANC< 1000/mm^3) with fever (a single temperature > 38.3°C or a sustained temperature of ≥ 38°C for more than 1 hour (h)), Grade ≥ 3 thrombocytopenia, Grade ≥ 2 bleeding (eg, gastrointestinal, respiratory, epistaxis, purpura), Grade ≥ 3 non hematologic toxicity, except- Grade 3 nausea or emesis with maximum duration of 48 h on adequate medical therapy and Grade 3 diarrhea which persists for < 72 h in the absence of maximal medical therapy, Grade ≥ 2 non hematologic treatment emergent adverse event (TEAE) that in the opinion of the investigator was of potential clinical significance such that further dose escalation would expose participants to unacceptable risk, treatment interruption ≥ 7 days due to unresolved toxicity.
Time Frame: Day 1 through Day 28
Population: The DLT Analysis Set included all participants in the Safety Analysis Set who completed all treatment and safety procedures through Day 28, inclusive, or experienced a DLT prior to Day 28, exclusive.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Phase 2 Dose Expansion: Non-progression Rate at Week 24 According to Prostate Cancer Working Group (PCWG2) Criteria
Description: The non-progression rate at Week 24 was defined as the proportion of participants who did not progress by Week 24.
Time Frame: Week 24
Population: The Phase 2 Dose Expansion of the study was not conducted.
Groups:
- Monotherapy: Alobresib 2 mg: Participants who had progressed on either abiraterone and/or enzalutamide, received alobresib 2 mg tablets administered orally once daily to determine the MTD.
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Phase 1b Dose Escalation: Cmax: Maximum Observed Plasma Concentration of Alobresib
Description: Cmax is the maximum observed concentration of drug in plasma.
Time Frame: Monotherapy: Predose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose on Cycle 1 Day 8 and Cycle 2 Day 1; Combination therapy: Predose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose on Cycle 1 Days 1 and 15
Population: The PK Analysis Set included participants who took at least 1 dose of study drug and have at least 1 non-missing postdose concentration value. Participants with available data were analyzed.
  Monotherapy: Samples were not collected at Cycle 1 Day 1 and Cycle 1 Day 15; samples were only collected for participants who received alobresib 3 mg, 6 mg and 9 mg doses at Cycle 2 Day 1. Combination Therapy: Samples were not collected at Cycle 1 Day 8 and Cycle 2 Day 1.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 6 | 2
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Cycle 1 Day 1 |  |  |  |  |  | 111.07 (37.957) | 199.00 (9.899)
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 4 | 3 | 6 | 4 | 0 | 0
  Cycle 1 Day 8 | 263.00 (141.875) | 263.75 (132.011) | 367.33 (49.359) | 293.33 (123.362) | 526.00 (280.391) |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 2
  Cycle 1 Day 15 |  |  |  |  |  | 84.4 (48.58) | 173.5 (28.99)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 1 | 0 | 0
  Cycle 2 Day 1 |  | 220.50 (95.459) |  | 203.50 (143.543) | 641.00 (NA) — Standard Deviation (SD) was not estimable for 1 participant. |  |

4. Secondary Outcome: Phase 1b Dose Escalation: Ctau: Observed Drug Concentration at the End of the Dosing Interval of Alobresib
Description: Ctau is the observed concentration of drug in plasma at the end of dosing.
Time Frame: Monotherapy: Predose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose on Cycle 1 Day 8 and Cycle 2 Day 1; Combination therapy: Predose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose on Cycle 1 Day 15
Population: Participants in the PK Analysis Set with available data were analyzed.
  Monotherapy: Samples were not collected at Cycle 1 Day 15; samples were only collected for participants who received alobresib 3 mg, 6 mg and 9 mg doses at Cycle 2 Day 1. Combination Therapy: Samples were not collected at Cycle 1 Day 8 and Cycle 2 Day 1.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 6 | 2
ng/mL
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 4 | 3 | 6 | 2 | 0 | 0
  Cycle 1 Day 8 | 180.00 (77.679) | 156.78 (100.307) | 141.67 (22.811) | 70.93 (32.905) | 157.20 (126.996) |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 2
  Cycle 1 Day 15 |  |  |  |  |  | 8.8 (7.77) | 3.9 (3.21)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 1 | 0 | 0
  Cycle 2 Day 1 |  | 127.60 (59.963) |  | 33.80 (NA) — SD was not estimable for 1 participant. | 268.00 (NA) — SD was not estimable for 1 participant. |  |

5. Secondary Outcome: Phase 1b Dose Escalation: AUClast: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Quantifiable Concentration of Alobresib
Description: AUClast is the concentration of drug over time zero to last concentration (area under the plasma concentration versus time curve).
Time Frame: as for outcome 3
Population: Participants in the PK Analysis Set with available data were analyzed.
  Monotherapy: Samples were not collected at Cycle 1 Day 1 and Cycle 1 Day 15; samples were only collected for participants who received alobresib 3 mg, 6 mg and 9 mg doses at Cycle 2 Day 1. Combination Therapy: Samples were not collected at Cycle 1 Day 8 and Cycle 2 Day 1.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 6 | 2
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Cycle 1 Day 1 |  |  |  |  |  | 1026.99 (359.220) | 1741.42 (737.521)
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 4 | 3 | 6 | 4 | 0 | 0
  Cycle 1 Day 8 | 4207.55 (2319.854) | 3742.30 (2106.308) | 4646.08 (890.441) | 3105.70 (1008.730) | 4494.79 (4124.948) |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 2
  Cycle 1 Day 15 |  |  |  |  |  | 652.7 (395.52) | 701.3 (353.25)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 1 | 0 | 0
  Cycle 2 Day 1 |  | 3264.79 (2024.141) |  | 1709.71 (264.402) | 10264.74 (NA) — SD was not estimable for 1 participant. |  |

6. Secondary Outcome: Phase 1b Dose Escalation: AUCtau: Area Under the Plasma Concentration Versus Time Curve Over the Dosing Interval of Alobresib
Description: AUCtau is defined as the concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 6 | 2
h*ng/mL
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 0 | 0
  Cycle 1 Day 8 | 4264.51 (2384.628) | 3758.92 (2076.013) | 4655.48 (949.099) | 3128.58 (998.059) | 7217.02 (4559.957) |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Cycle 1 Day 15 |  |  |  |  |  | 765.3 (373.39) | 701.3 (353.25)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 1 | 0 | 0
  Cycle 2 Day 1 |  | 3243.01 (2110.324) |  | 1522.75 (NA) — SD was not estimable for 1 participant. | 10264.74 (NA) — SD was not estimable for 1 participant. |  |

7. Secondary Outcome: Phase 1b Dose Escalation: Tmax: Time (Observed Time Point) of Cmax of Alobresib
Description: Tmax is the time observed for the Cmax of alobresib.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 6 | 2
hours
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Cycle 1 Day 1 |  |  |  |  |  | 1.07 [0.50 to 2.92] | 0.46 [0.42 to 0.50]
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 0 | 0
  Cycle 1 Day 8 | 0.50 [0.48 to 23.85] | 0.66 [0.50 to 1.05] | 0.58 [0.50 to 2.00] | 1.42 [0.50 to 3.97] | 0.72 [0.50 to 2.08] |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 2
  Cycle 1 Day 15 |  |  |  |  |  | 0.5 [0.5 to 7.9] | 0.5 [0.5 to 0.5]
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 1 | 0 | 0
  Cycle 2 Day 1 |  | 1.76 [0.50 to 3.02] |  | 4.93 [3.87 to 6.00] | 4.08 [4.08 to 4.08] |  |

8. Secondary Outcome: Percentage of Participants Who Had ≥ 30% Reduction in Prostate Specific Antigen (PSA) From Baseline at Week 12
Description: PSA response was defined as percentage of participants with ≥ 30% decline in PSA from baseline by 12 weeks.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 6 | 2
percentage of participants | 0.0 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0

9. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the interval from first dose date of study drug to the earlier of the first documentation of definitive disease progression (assessed per PCWG2) or death from any cause. PCWG2 criteria for progression was determined as 'Decline from baseline' when record start of therapy to first prostate-specific antigen (PSA) increase that is ≥ 25% and ≥ 2 ng/mL above the nadir and confirmed by a second value 3 or more weeks later; 'No decline from baseline' when PSA progression ≥ 25% and ≥ 2 ng/mL after 12 weeks.
Time Frame: Up to approximately 4 years
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 4 | 3 | 2 | 6 | 4 | 5 | 1
months | 2.61 [1.58 to 8.61] | 2.10 [1.97 to 2.60] | 4.17 [2.79 to 5.55] | 2.78 [2.69 to 11.07] | 2.69 [0.53 to 14.00] | 3.25 [1.15 to 21.59] | 5.98 [NA to NA] — Upper and lower limit of 95% confidence interval are not estimable for 1 participant.

10. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval from first dose date of study drug to death from any cause.
Time Frame: Up to approximately 4 years
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 5 | 6 | 2
months | NA [NA to NA] — Data were not evaluable because participants discontinued the study without death. | NA [3.12 to NA] — Data were not evaluable because participants discontinued the study without death. | NA [NA to NA] — Data were not evaluable because participants discontinued the study without death. | NA [NA to NA] — Data were not evaluable because participants discontinued the study without death. | NA [NA to NA] — Data were not evaluable because participants discontinued the study without death. | NA [1.15 to NA] — Data were not evaluable because participants discontinued the study without death. | NA [NA to NA] — Data were not evaluable because participants discontinued the study without death.

ADVERSE EVENTS:
Time Frame: Adverse Events: From first dose through last dose of the study drug (maximum: 131 weeks) plus 30 days; All-Cause Mortality: First dose date up to approximately 4 years
Description: The Safety Analysis Set included all participants who received >= 1 dose of study treatment with treatment group designated according to actual treatment.
Arm/Group | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Monotherapy: Alobresib 9 mg | Combination Therapy: Alobresib 3 mg + Enzalutamide | Combination Therapy: Alobresib 6 mg + Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/4 | 0/3 | 0/6 | 0/5 | 1/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/4 | 1/3 | 1/6 | 2/5 | 2/6 | 1/2
Other Adverse Events (participants affected / at risk) | 5/5 | 3/4 | 3/3 | 6/6 | 5/5 | 5/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: Alobresib 2 mg (N=5) | Monotherapy: Alobresib 3 mg (N=4) | Monotherapy: Alobresib 4 mg (N=3) | Monotherapy: Alobresib 6 mg (N=6) | Monotherapy: Alobresib 9 mg (N=5) | Combination Therapy: Alobresib 3 mg + Enzalutamide (N=6) | Combination Therapy: Alobresib 6 mg + Enzalutamide (N=2)
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: Alobresib 2 mg (N=5) | Monotherapy: Alobresib 3 mg (N=4) | Monotherapy: Alobresib 4 mg (N=3) | Monotherapy: Alobresib 6 mg (N=6) | Monotherapy: Alobresib 9 mg (N=5) | Combination Therapy: Alobresib 3 mg + Enzalutamide (N=6) | Combination Therapy: Alobresib 6 mg + Enzalutamide (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 2 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site extravasation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Device related thrombosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 3 | 3 | 4 | 2 | 1
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 4 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or The study has been completed at all study sites for at least 2 years.

DOCUMENTS (2):
  • Study Protocol (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT02607228/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT02607228/SAP_001.pdf